CLINICAL TRIAL: NCT06295471
Title: A Comparative Clinical Study to Assess Pain Score and Wound Healing Following Fractional Ablation With a Difference Frequency Generation (DFG) Laser and Carbon Dioxide (CO2) Laser
Brief Title: A Comparative Clinical Study to Assess Pain Score and Wound Healing Following Fractional Ablation With a DFG Laser and CO2 Laser
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Dieter Manstein, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2024P000112
Record Dates: First submitted 2024-02-21; First posted 2024-03-06 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Healthy
Keywords: Laser
MeSH Terms: interventions — Lasers, Gas; Tomography, Optical Coherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Treatment (Experimental): 23 healthy subjects with treatment of the DFG and CO2 laser
  Interventions: Device: DFG Laser; Device: CO2 Laser; Device: Optical coherence tomography (OCT)

INTERVENTIONS:
Device: DFG Laser — Laser treatment to the upper thigh
Device: CO2 Laser — Laser treatment to the upper thigh
Device: Optical coherence tomography (OCT) — Angiographic OCT imaging at areas of interest

SUMMARY:
This research study aims assess whether the Difference Frequency Generation (DFG) laser could be a better alternative to the CO2 laser in terms of reduced side effects and patient downtime.

DETAILED DESCRIPTION:
The primary goal of this study is to compare the pain score and wound healing time in healthy subjects undergoing low fluence fractional ablation using the DFG and CO2 lasers. The secondary objective involves assessing the impact of each laser on dermal vasculature using an Optical Coherence Tomography (OCT) imaging system.

Participants will be treated with the DFG and CO2 laser to the upper thighs. Photography, pain scores, and OCT imaging will be recorded over the course of the study visits.

The investigators plan to enroll 23 healthy subjects to complete the study. Subjects must be equal to greater than 18 years old and may be any gender or Fitzpatrick skin type.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be able and willing to provide written informed consent and comply with the requirements of the study protocol;
* Subjects must be in good general health, based on answers provided during the screening visit;
* Subjects must be able to read and understand English.
* Subjects must be above the age of 18.
* Subjects must have no history of skin conditions that affect the integrity of the skin barrier.

Exclusion Criteria:

* Are pregnant or lactating;
* Have a history of drug or alcohol abuse or have reported habitual alcohol intake greater than 2 standard drinks per day [e.g., 2 beers, 2 glasses of wine, or 2 mixed drinks];
* Are smoking or have a history of smoking;
* Presence of eczema, psoriasis, skin wounds or ulcers, or any other skin disease on the thighs;
* Have birth marks, tattoos, scars, or any other disfiguration of the skin in the skin area of interest;
* Presence of sunburn or tan in the treatment area;
* Use of any topical application of retinoids in the area of interest or systemic retinoids in the past 6 months;
* Use of any prescription topical medication, such as corticosteroids or hydroquinone on the skin area of interest in the past 6 months;
* History of blood-clotting abnormality;
* History of keloid formation or hypertrophic scarring;
* History of allergic reaction to local anesthesia, aluminum chloride, and/or glycerol;
* Investigator, interfere with study evaluations or pose a risk to subject safety during the study;
* Exhibits any clinical conditions or takes any medication which in the opinion of the investigator may interfere with the study or pose a risk to subject safety during the study;
* Is not able to follow study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2024-10-16 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) pain score | 90 minutes
  Subjects will report pain score using VAS for the CO2 and DFG laser treated areas at Visit 1. The VAS is a 10cm long scale with 0cm representing "no pain" and 10cm representing "worst possible pain".
Wound healing time | 1 month
  Wound healing of the laser treated areas will be assessed and compared via photography at each visit.

SECONDARY OUTCOMES:
Vessel density via OCT imaging | 1 month
  The OCT system will be used to assess re-epithelialization and dermal vasculature of laser treated areas at each visit
Vessel length via OCT imaging | 1 month
  The OCT system will be used to assess re-epithelialization and dermal vasculature of laser treated areas at each visit
Vessel thickness via OCT imaging | 1 month
  The OCT system will be used to assess re-epithelialization and dermal vasculature of laser treated areas at each visit

CONTACTS AND LOCATIONS:
Overall Officials: Dieter Manstein, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- MGH Clinical Unit for Research Trials & Outcomes in Skin, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data (IPD) available to other researchers.

REFERENCES:
- [Background] Ibrahim O, Wenande E, Hogan S, Arndt KA, Haedersdal M, Dover JS. Challenges to laser-assisted drug delivery: Applying theory to clinical practice. Lasers Surg Med. 2018 Jan;50(1):20-27. doi: 10.1002/lsm.22769. Epub 2017 Nov 20. PMID 29154501
- [Background] Ko DY, Kim KH, Song KH. A randomized trial comparing methyl aminolaevulinate photodynamic therapy with and without Er:YAG ablative fractional laser treatment in Asian patients with lower extremity Bowen disease: results from a 12-month follow-up. Br J Dermatol. 2014 Jan;170(1):165-72. doi: 10.1111/bjd.12627. PMID 24102369
- [Background] Haak CS, Togsverd-Bo K, Thaysen-Petersen D, Wulf HC, Paasch U, Anderson RR, Haedersdal M. Fractional laser-mediated photodynamic therapy of high-risk basal cell carcinomas--a randomized clinical trial. Br J Dermatol. 2015 Jan;172(1):215-22. doi: 10.1111/bjd.13166. Epub 2014 Nov 30. PMID 24903544
- [Background] Togsverd-Bo K, Haak CS, Thaysen-Petersen D, Wulf HC, Anderson RR, Haedersdal M. Intensified photodynamic therapy of actinic keratoses with fractional CO2 laser: a randomized clinical trial. Br J Dermatol. 2012 Jun;166(6):1262-9. doi: 10.1111/j.1365-2133.2012.10893.x. PMID 22348388
- [Background] Waibel JS, Wulkan AJ, Shumaker PR. Treatment of hypertrophic scars using laser and laser assisted corticosteroid delivery. Lasers Surg Med. 2013 Mar;45(3):135-40. doi: 10.1002/lsm.22120. Epub 2013 Mar 4. PMID 23460557
- [Background] Choi SH, Kim KH, Song KH. Efficacy of ablative fractional laser-assisted photodynamic therapy with short-incubation time for the treatment of facial and scalp actinic keratosis: 12-month follow-up results of a randomized, prospective, comparative trial. J Eur Acad Dermatol Venereol. 2015 Aug;29(8):1598-605. doi: 10.1111/jdv.12953. Epub 2015 Feb 1. PMID 25640401
- [Background] Haedersdal M, Sakamoto FH, Farinelli WA, Doukas AG, Tam J, Anderson RR. Fractional CO(2) laser-assisted drug delivery. Lasers Surg Med. 2010 Feb;42(2):113-22. doi: 10.1002/lsm.20860. PMID 20166154
- [Background] Manstein D, Herron GS, Sink RK, Tanner H, Anderson RR. Fractional photothermolysis: a new concept for cutaneous remodeling using microscopic patterns of thermal injury. Lasers Surg Med. 2004;34(5):426-38. doi: 10.1002/lsm.20048. PMID 15216537
- [Background] Chen KH, Tam KW, Chen IF, Huang SK, Tzeng PC, Wang HJ, Chen CC. A systematic review of comparative studies of CO2 and erbium:YAG lasers in resurfacing facial rhytides (wrinkles). J Cosmet Laser Ther. 2017 Aug;19(4):199-204. doi: 10.1080/14764172.2017.1288261. Epub 2017 Feb 6. PMID 28166434
- [Background] Ross EV, Swann M, Soon S, Izadpanah A, Barnette D, Davenport S. Full-face treatments with the 2790-nm erbium:YSGG laser system. J Drugs Dermatol. 2009 Mar;8(3):248-52. PMID 19271372
- [Background] Weinstein C. Erbium laser resurfacing: current concepts. Plast Reconstr Surg. 1999 Feb;103(2):602-16; discussion 617-8. doi: 10.1097/00006534-199902000-00038. PMID 9950553
- [Background] Wang-Evers M, Blazon-Brown AJ, Ha-Wissel L, Arkhipova V, Paithankar D, Yaroslavsky IV, Altshuler G, Manstein D. Assessment of a 3050/3200 nm fiber laser system for ablative fractional laser treatments in dermatology. Lasers Surg Med. 2022 Aug;54(6):851-860. doi: 10.1002/lsm.23550. Epub 2022 Apr 8. PMID 35395696
- [Background] Lv K, Liu H, Xu H, Wang C, Zhu S, Lou X, Luo P, Xiao S, Xia Z. Ablative fractional CO2 laser surgery improving sleep quality, pain and pruritus in adult hypertrophic scar patients: a prospective cohort study. Burns Trauma. 2021 Jul 27;9:tkab023. doi: 10.1093/burnst/tkab023. eCollection 2021. PMID 34322556